CLINICAL TRIAL: NCT02889705
Title: Longitudinal Follow-up of Muscle Echotextures in Infants With Congenital Muscular Torticollis
Brief Title: Echotexture in Following Muscle Fibrosis
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Chih-Chin Hsu, Doctor, Chang Gung Memorial Hospital
Other Study IDs: 100-4436B
Record Dates: First submitted 2016-08-26; First posted 2016-09-05 (Estimated); Last update posted 2016-09-05 (Estimated); Status verified 2016-08

CONDITIONS: Congenital Muscular Torticollis
Keywords: Ultrasonography; echotexture; K value; SCM muscles; CMT infants
MeSH Terms: conditions — Congenital torticollis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Other: Ultrasonographic examination

SUMMARY:
Objective: To document the sternocleidomastoid (SCM) muscle fibrosis in congenital muscular torticollis (CMT) infants with quantified echotexture and measured thickness during the treatment course.

Design: Cohort study. Setting: Rehabilitation department in a tertiary care hospital. Participants: Infants with clinical diagnosis of CMT, without any neurological presentation, cervical spin abnormality, and developmental dysplastic hip problem, were recruited in the study.

Intervention: All subjects had physiotherapy for at least 3 months. They underwent at least two times of clinical assessment and ultrasonographic examination (1) for bilateral SCM muscles during the follow-up period.

End of follow-up: Subjects who still had prominent clinical presentations after physiotherapy for 6 months or were older than 1 year would receive surgery. Subsided presenting clinical features determined by the clinician was the other end-point of this investigation.

Main Outcome Measures: The K value, derived from the difference of echo intensities (2) between the involved and uninvolved SCM muscles on longitudinal sonograms, was used to represent the severity of muscle fibrosis in CMT infants. Bilateral SCM muscle thickness and involved-to-uninvolved thickness ratio (Ratio I/U) were also obtained from longitudinal sonograms. Clinical outcome was also recorded.

DETAILED DESCRIPTION:
1. An experienced sonographer performed ultrasonographic examination with the subject in the supine position and heads rotated contralaterally to the examination side. A 5-12 MHz linear-array ultrasound transducer was used to observe both longitudinal and transverse views of bilateral SCM muscles for each subject. The ultrasound system settings, including gain (86%), monitor dynamic range (70 dB), and depth (2 cm), were kept constant throughout the study.
2. The echo intensity was determined by computer-assisted gray scale analysis and was calculated in MATLAB 2006b. The mean echo intensity of every pixel in the region of interest and the K value developed to compare sonograms between different individuals or between different times in the same subject were estimated as the previous study (PMID: 22215768)

ELIGIBILITY:
Inclusion Criteria:

* infants with congenital muscular torticollis Presenting clinical features of the CMT infants, including head tilt in the upright position, facial asymmetry, limited passive range of motion in neck rotation, palpable neck mass

Exclusion Criteria:

* Subjects with neurological symptoms or signs
* Cervical spine abnormalities
* Developmental dysplastic hip problems

Ages: 1 Month to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Convenience sample of infants in both gender with congenital muscular torticollis, are reviewed by the exclusion criteria (please see below). Subjects, whose parents are willing to sign the informed consent and fit our inclusion/exclusion criteria are prospectively enrolled in this study.
  Age, gender distribution, body weight (BW), body length (BL), affected muscle side, follow-up period, and interval between two visits were also recorded.
  Physiotherapy of passive stretching of the involved muscle, positioning, and massage were capable of diminishing the development of scoliosis and facial asymmetry in the future.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2012-08; Primary Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
K value | 3 years
  Difference of echo intensities on muscle sonograms between involved and uninvolved sternocleidomastoid muscles in 50 infants with congenital muscular torticollis
Muscle thickness in cm | 3 years
  Bilateral sternocleidomastoid muscle thickness in 50 infants with congenital muscular torticollis
Ratio I/U (involved-to-uninvolved muscle thickness ratio) | 3 years
Age in month | 3 years
  The age of first evaluation
Times of ultrasonographic examinations | 3 years
  The times of ultrasonographic examination before end follow-up
Body weight in kg | 3 years
  Body weight of all subjects during the follow-up period
Body length in cm | 3 years
  Body length of all subjects during the follow-up period